CLINICAL TRIAL: NCT02816619
Title: Evaluation of a Personalized Physical Activity Coaching Program in Parkinson's Disease
Acronym: APA-PARK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Laboratoire des Adaptations Métaboliques à l'Exercice en conditions Physiologiques et Pathologiques (Other); UFR STAPS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHU-0265; 2016-A00040-51 (Registry Identifier: 2016-A00040-51)
Record Dates: First submitted 2016-06-03; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Physical activity; Physical exercise
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- APA+ (Experimental): APA + : patients will beneficiate of Personalized Physical Activity coaching program during 3 months (1 hour, twice by week, during 3 months)
  Interventions: Behavioral: Personalized Physical Activity coaching program
- APA- (Other): APA- : patients will do free practice of physical activity during 3 months.
  Interventions: Behavioral: Free practice of physical activity

INTERVENTIONS:
Behavioral: Personalized Physical Activity coaching program
  Arms: APA+
Behavioral: Free practice of physical activity
  Arms: APA-

SUMMARY:
There is growing interest for physical activity in Parkinson's disease in order to improve mobility and function of these patients. It seems from previous studies that difficulty, intensity and specificity of physical exercises are important parameters conditioning the effect of physical activity on cerebral plasticity and clinical improvement.

Thus, the aim of this study is to evaluate the benefits of a Personalized Physical Activity coaching program, including scheduled and frequent follow up associated with progressive readaptation of exercise intensity depending on individual performances (during 3 months), versus free practice of physical activity in Parkinson's disease.

DETAILED DESCRIPTION:
Type of study: a randomized, single-blind, parallel-group, controlled clinical trial.

Number of centers: 1 (Clermont-Ferrand)

Patients

Patients eligible for inclusion will be randomized to one of the two groups:

* APA + : patients will beneficiate of Personalized Physical Activity coaching program during 3 months (1 hour, twice by week, during 3 months)
* APA- : patients will do free practice of physical activity during 3 months.

Study Performance Patients will be evaluated 3 times : at J0 (baseline, V1), 3 months after Personalized Physical Activity coaching program (J0+3M, V2), and 3 months after the end of the Personalized Physical Activity coaching program (J0+6M)

V1:

* Signature of an informed consent form.
* Demographic and clinical characteristics (sex, age, disease duration, treatments).

V1, V2, V3

* Neurological evaluation (Unified Parkinson Disease Rating Scale part III score)
* Evaluation of quality of life (Parkinson's Disease Questionnaire 39-item version (PDQ-39), participation to Daily life activities (Lawton and Brody Activities of Daily Living scale (IADL questionnaire25)
* Evaluation of performances for specific tests for balance (stabilometry), muscular strength (isometry)
* Evaluation of cardiorespiratory function (VO2pic et 6 min Walk Test)
* Evaluation of body composition (lean body mass/fat mass) with DEXA.
* Dropout rates at V2 and V3
* Evaluation of the activity with the eMOUVE application in a subgroup of patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical criteria for Parkinson's disease
* Men or women aged from 18 to 80 years old.
* Social security coverage.
* Ability to provide informed consent.

Exclusion Criteria:

* neurological disease other than Parkinson's disease
* severe depression (Beck Depression Inventory>37) or psychiatric comorbidities (UPDRS I )
* significant cognitive impairment (MoCA<24)
* orthopedic impairment with functional restriction
* contraindication to physical exercise

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-06 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of the Unified Parkinson Disease Rating Scale part III score | at +3months

SECONDARY OUTCOMES:
Change from baseline of Parkinson's Disease Questionnaire 39-item version score | at +3months
Change from baseline of the Lawton and Brody Activities of Daily Living scale score | at +3months
Change from baseline of the percentage of sedentarity, mild, moderate and intense activity using the eMOUVE application | at +3months
Change from baseline of percentage of sedentarity, mild, moderate and intense activity using the eMOUVE application | at + 6 months
Change from baseline of balancing abilities measured by stabilometry | at +3months
Change from baseline of balancing abilities measured by stabilometry | at + 6 months
Change from baseline of muscular strength measured with isometric test | at +3months
Change from baseline of muscular strength measured with isometric test | at +6months
Change from baseline of VO2pic | at +3months
Change from baseline of VO2pic | at + 6 months
Change from baseline of the 6 min Walking Test score | at +3 months
Change from baseline of the 6 min Walking Test score | at + 6 months
Change from baseline of fat and lean body mass measured by DEXA | at +3 months.
Change from baseline fat and lean body mass measured by DEXA | at +6 months.
dropout rates | at +3 months
dropout rates | at +6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Zanchet C, Lambert C, Boyer T, Pereira B, Derost P, Debilly B, Duclos M, Boisseau N, Marques A. Effect of an adapted physical activity program in Parkinson's disease: A randomized controlled study (APA-Park). Parkinsonism Relat Disord. 2025 May;134:107777. doi: 10.1016/j.parkreldis.2025.107777. Epub 2025 Mar 10. PMID 40088781
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886